CLINICAL TRIAL: NCT00323271
Title: Cognitive-behavior Therapy for MS-Related Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D4150-R
Record Dates: First submitted 2006-05-05; First posted 2006-05-09 (Estimated); Results first posted 2015-09-25 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-08

CONDITIONS: Multiple Sclerosis
Keywords: Chronic pain; Cognitive behavioral therapy; Multiple sclerosis; Randomized controlled trial
MeSH Terms: conditions — Multiple Sclerosis; Chronic Pain | interventions — Cognitive Behavioral Therapy; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Behavioral: Cognitive-behavior therapy
  Interventions: Behavioral: Cognitive-behavior therapy
- Arm 2 (Active Comparator): Interventional: Educational intervention
  Interventions: Other: Interventional

INTERVENTIONS:
Behavioral: Cognitive-behavior therapy — CBT: The components of CBT include (1) identification of idiosyncratic beliefs about pain and pain treatment, as well as reconceptualization of the pain experience as subject to personal control (sessions 1-2), (2) instruction in specific cognitive (e.g., distraction) and behavioral (e.g., change in activity patterns such as alternating activity with periods of rest) skills (sessions 3-8), and (3) consolidation of cognitive/behavioral skills through activities such as role playing (sessions 9-11).
  Arms: Arm 1
Other: Interventional — Educational intervention: Session topics will include information on the etiology of MS, MS subtypes and disease progression, common symptoms of MS, medical management of MS, rehabilitation approaches to management of MS-related symptoms, exercise, sick day management, stress management, psychosocial adjustment, family involvement, and appropriate use of the health care system.
  Arms: Arm 2

SUMMARY:
The purpose of this study is to evaluate the efficacy of a brief psychological intervention, cognitive-behavior therapy, for the management of persistent pain associated with Multiple Sclerosis.

DETAILED DESCRIPTION:
The primary purpose of the proposed study is to evaluate the feasibility and efficacy of tailored CBT with standard pharmaceutical care (CBT/SC) in reducing pain, disability, and distress among persons with Multiple Sclerosis (MS) related pain conditions. This will entail: (1) evaluating the feasibility, perceived credibility, participation and adherence rates, and satisfaction related to CBT, (2) conducting a randomized controlled trial of the efficacy of CBT relative to an education control/standard care (ED/SC) condition, and (3) evaluating possible predictors of treatment response including demographics, disease-relevant variables, cognitive functioning, and motivation or readiness to adopt a self-management approach to MS-related pain.

Research Design: A randomized mixed factorial controlled design will be employed in which CBT/SC is compared to EDSC. Repeated assessments of key outcome domains will occur at pretreatment/baseline, at 15 weeks (post-treatment), and 20, 36, and 52 (follow-up) weeks.

Methodology: Participants in this trial will be 124 persons with MS (including veterans and non-veterans) who report persistent MS-related pain (e.g., neuropathic pain, pain related to muscle spasms, neuralgias) of at least moderate intensity (pain severity of 4 or greater on the numeric rating scale) despite optimal pharmacological management. Participants must be at least 21 years of age and able to provide informed consent. Exclusion criteria include: (1) pending surgery or interventional anesthesiological procedures for pain, (2) currently psychotic or actively suicidal or homicidal, (3) current alcohol or substance abuse or dependence, (4) presence of other life threatening illnesses, (5) the presence of profound cognitive impairment rendering successful participation in CBT or ED impossible, (6) the presence of physical disabilities resulting in an inability to attend treatment sessions and/or inability to participate in telephone interventions (e.g., severe dysarthria), (7) prior or current psychological treatment for chronic pain, (8) two or more documented exacerbations of MS-related symptoms during the past year, and (9) current exacerbation of symptoms defined as sudden onset of symptoms within a 24 hour period. CBT will involve an innovative treatment approach that combines specific training in relevant cognitive and behavior skills targeting management of pain and the negative impacts of pain. The application of these skills for the management of coincident symptoms of MS (e.g., spasticity, fatigue, abnormal sensory experiences) will also be encouraged. ED will involve provision of a broad array of educational material regarding MS and its management, but it will not explicitly inform participants about non-pharmacological strategies for management of pain. Both treatments will involve seven 60 minute, outpatient individual treatment sessions offered every other week, interspersed with five, 30 minute individual telephone sessions (one final face-to-face session will be 30 minute individual telephone sessions will be included) provided by a psychologist and supported by patient education and treatment guides that have been developed for the study. Participants will be randomly assigned to one of two treatment arms: CBT/SC or ED/SC. Recruitment rates, session adherence, dropout rates, and participants' ratings of comprehension, treatment credibility, treatment satisfaction and adherence to therapist recommendations will be used to assess feasibility of the treatment and recruitment methods. Multiple standardized measures of each outcome domain of interest will be obtained, including pain severity, disability, affective distress, and quality of life. The analysis of each of the primary and secondary outcome measures (summary measures of pain intensity, pain-related disability, MS-related disability, and emotional functioning) will be by a repeated measures mixed effects model27. The outcome variable in each model will be the changes at each follow-up visit relative to baseline, with the baseline value included as a covariate in the model. Several possible predictors of treatment adherence and outcome will be examined, including participant demographics (e.g., age, gender, ethnicity), disease-relevant variables (e.g.., MS subtype, disease duration, disease severity, level of cognitive functioning), outcome measures (e.g., pain severity, depressive symptom severity), and a measure of motivation for adoption of a self-management approach to chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* a confirmed diagnosis of Multiple Sclerosis,
* history of daily pain or discomfort (burning, tingling or other parenthesis) for a period of 3 months immediately prior to enrollment,
* judgment of one of the study neurologists (AL or MK) that the pain reported by the patient is either directly [e.g., pain associated with optic neuritis and neuralgias] or indirectly related [e.g., pain due to painful muscle contractures and spasms] to MS and/or its treatment (persons with pain that is judged to be entirely coincident with MS [e.g., idiopathic low back pain] will not be included),
* documentation of optimal pharmacological management of MS-related pain and confirmation of this judgment by one of the study neurologists,
* continued use of appropriate pharmaceuticals for the management of MS and pain, and
* continued refractory pain despite pharmaceutical intervention as described above (as determined by a pain intensity score 4 on a 0-10 numeric rating scale).

Exclusion Criteria:

* pending surgery or interventional anesthesiological procedures for pain,
* currently psychotic or actively suicidal or homicidal,
* current alcohol or substance abuse or dependence,
* presence of other life threatening illnesses,
* the presence of profound cognitive impairment rendering successful participation in CBT or ED impossible,
* the presence of physical disabilities resulting in an inability to attend treatment sessions and/or inability to participate in telephone interventions (e.g., severe dysarthria),
* prior or current psychological treatment for chronic pain,
* two or more documented exacerbations of MS-related symptoms during the past year, and
* current exacerbation of symptoms defined as sudden onset of symptoms within a 24 hour period. Participants experiencing an exacerbation will be included after a one-month period of appropriate treatment or three months after the onset of the exacerbation. The Exacerbation Questionnaire, also described below and developed by Dr. Mohr, one of our co-investigators, will be used to assess and monitor significant exacerbations of MS. The Multiple Sclerosis Functional Composite (MSFC) score described below will be used to determine these later two exclusion criteria.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2006-07; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert D. Kerns, PhD, Principal Investigator — VA Connecticut Health Care System (West Haven)
Locations (2):
- United States (2):
  - VA Connecticut Health Care System (West Haven), West Haven, Connecticut
  - VA Medical Center, Jamaica Plain Campus, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occured during April 2007 through September 2009.
  Participants were Veterans and nonVeterans recruited primarily through their providers in one of three treatment settings, namely the MS Clinics at the VA Connecticut Healthcare System and VA Boston Healthcare System and at the Yale MS Center.
Pre-assignment Details: 1 subject enrolled into the study but was found to be ineligible before randomization.
Groups:
- Cognitive-behavior Therapy: Behavioral: Cognitive-behavior therapy
  Cognitive-behavior therapy: CBT: The components of CBT include (1) identification of idiosyncratic beliefs about pain and pain treatment, as well as reconceptualization of the pain experience as subject to personal control (sessions 1-2), (2) instruction in specific cognitive (e.g., distraction) and behavioral (e.g., change in activity patterns such as alternating activity with periods of rest) skills (sessions 3-8), and (3) consolidation of cognitive/behavioral skills through activities such as role playing (sessions 9-11).
- Educational Intervention: Interventional: Educational intervention
  Interventional: Educational intervention: Session topics will include information on the etiology of MS, MS subtypes and disease progression, common symptoms of MS, medical management of MS, rehabilitation approaches to management of MS-related symptoms, exercise, sick day management, stress management, psychosocial adjustment, family involvement, and appropriate use of the health care system.
Period: Overall Study
Arm/Group | Cognitive-behavior Therapy | Educational Intervention
Started | 13 | 12
Completed | 11 | 9
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive-behavior Therapy | Educational Intervention | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.23 (8.691) | 54.67 (12.361) | 53.95 (10.408)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 8 | 8 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 10 | 10 | 20
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity
Description: The Numeric Rating Scale of pain intensity (NRS-I) is an 11-point numeric rating scale (0 = no pain, 10 = worst pain imaginable). Participants were asked to rate their usual, worst and least pain over the past week. The average of these numbers will serve as the primary outcome measure.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive-behavior Therapy | Educational Intervention
Number analyzed (Participants) | 13 | 12
units on a scale | 5.31 (2.213) | 5.42 (2.610)
Statistical Analysis 1: Comparison: Cognitive-behavior Therapy vs Educational Intervention; Test type: Superiority or Other; p = .911, t-test, 2 sided; Mean Difference (Final Values) = -0.108, 95% CI 2-sided [-2.106 to 1.888]

2. Primary Outcome: Pain Intensity
Description: as for outcome 1
Time Frame: Baseline to Post Treatment (12 weeks)
Population: Multiple imputation used to account for missing variables; pre-treatment rating and years of MS pain were covariates
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive-behavior Therapy | Educational Intervention
Number analyzed (Participants) | 13 | 12
units on a scale | 5.76 (1.53) | 5.12 (2.51)
Statistical Analysis 1: Comparison: Cognitive-behavior Therapy vs Educational Intervention; Test type: Superiority or Other; p = 0.320, ANCOVA — Multiple imputation used to account for missing variables; pre-treatment rating and years of MS pain were covariates; Mean Difference (Final Values) = 0.644, 95% CI 2-sided [-1.058 to 2.345]

ADVERSE EVENTS:
Time Frame: AEs and SAEs did not occur but participants were asked during each visit with the therapist and during each follow up. Recruitment timeframe was April 2007 to September 2009.
Arm/Group | Cognitive-behavior Therapy | Educational Intervention
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 0/13 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No